CLINICAL TRIAL: NCT04320810
Title: Developing Metagenomic Approaches to Identify the Causes of Pediatric Infectious Diseases
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: CHFudanU_NNICU13
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Infectious Disease
Keywords: Metagenome next generation sequencing; Pediatric
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mNGS diagnosis: Using mNGS to diagnosis infectious disease of this group
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — It's only observational study. No interventions.

SUMMARY:
Infectious diseases remain leading causes of mortality and morbidity in children. Rapid and accurate diagnosis of infectious diseases in children is important for developing an effective treatment and management strategy. However, the current diagnosis of infectious agents mainly depends on culture and molecular testing. Both of the methods either has long turnaround times or narrow detection range. Metagenome next generation sequencing (mNGS) has been applied to the diagnosis of central nervous system infection, lower respiratory tract infection and sepsis, which showed high positive rate, short turnaround time. However, there is currently no assessment of the diagnostic efficacy of mNGS in children infectious diseases. This study used the DNA extraction and library construction technology developed for children's low volume clinical samples to assess the sensitivity and specificity of mNGS in the diagnosis of infectious diseases, and the treatment outcome based on mNGS test results.

ELIGIBILITY:
Inclusion Criteria:

* Patients are highly suspected of sepsis；
* Patients are highly suspected of respiratory infections；
* Patients are highly suspected of central nervous system infection；
* Patients are highly suspected of fever of unknown origin

Exclusion Criteria:

* Congenital malformations；
* Patients requiring surgical intervention;
* Patients with skin barrier dysfunction

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study mainly focus on the pediatric patients who is suspected of infectious disease.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of metagenome next generation sequencing in the diagnosis of pediatric infectious disease | From the date of first samples enrolled until the last samples detected, up to 3 years
  Samples from patients, who is suspected to central nervous system infection, respiratory infection, bloodstream infection and other unknown infections, will be tested by mNGS and traditional methods simultaneously. The sensitivity value will be calculated by comparing the detecting results of mNGS and traditional detecting methods.
The specificity of metagenome next generation sequencing in the diagnosis of pediatric infectious disease | From the date of first samples enrolled until the last samples detected, up to 3 years
  Samples from patients, who is suspected to central nervous system infection, respiratory infection, bloodstream infection and other unknown infections, will be tested by mNGS and traditional methods simultaneously. The specificity value will be calculated by comparing the detecting results of mNGS and traditional detecting methods.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhou, Doctor, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China